CLINICAL TRIAL: NCT02612883
Title: Flux Measurement and Outcome in Major Abdominal Surgery
Acronym: FLUX
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Other Study IDs: VTG-04
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Perfusion
Keywords: Flux measurement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Esophagus: Measuring of tissue perfusion of the esophagus
- Liver: Measuring of tissue perfusion of the liver
- Stomach: Measuring of tissue perfusion of the stomach
- Pancreas: Measuring of tissue perfusion of the pancreas
- Colon: Measuring of tissue perfusion of the colon

SUMMARY:
Tissue perfusion is a critical factor for tissue regeneration and healing of anastomoses. Compromised microperfusion in the area where the anastomosis is sited likely contributes to leaks, but until now there has not been an easy and reliable technique to intraoperatively evaluate microperfusion.

Objectives: To assess the association of intraoperative flux measurement with postoperative outcome of patients undergoing major abdominal surgery.

Trial design: Prospective observational study. Flux measurement will be carried out using the moorVMS-LDF DUAL CHANNEL Laser Doppler Blood Flow system. The flux probe will be applied on the respective organs (i.e. esophagus, stomach, liver, pancreas, colon, rectum) and measurements will be documented after a stable signal has been obtained.

DETAILED DESCRIPTION:
Surgical resection is the primary therapy for a variety of benign and malignant diseases of the gastrointestinal tract. Advances in the perioperative care surgical technique and imaging modalities have significantly improved the outcome of patients with major abdominal resections within the past three decades. However, the incidence of postoperative complications after major abdominal resections remains high with morbidity rates of 30-60% despite a gradual decrease in perioperative mortality over time. Persistently high morbidity rates may in part be explained by broadened indications with surgery in patients having relevant comorbidities and/or advanced disease requiring extended resections. The reduction of perioperative morbidity is of high relevance for the patients, as complications are associated with poor oncological and functional long-term outcome and delay of further therapy. In addition, complications present a major cause of costs for the health care system.

Tissue perfusion is a critical factor for tissue regeneration and healing of anastomoses. Compromised microperfusion in the area where the anastomosis is sited likely contributes to leaks, but until now there has not been an easy and reliable technique to intraoperatively evaluate microperfusion.

During the post-operative period, inadequate wound perfusion and impairment of systemic or local oxygenation represent the main predisposing factors for anastomotic leakage. This is the case for the gastric conduit as well as for colonic/rectal anstomoses.

For example, the performance of gastroplasty has been shown to be associated with impairment in the microcirculatory blood flow in the proximal end of the gastric tube, despite the absence of significant impairment in systemic haemodynamic status.

These microcirculatory impairments promote the occurrence of oesophageal anastomotic leakage, which represents a potentially life-threatening complication related to the disastrous consequences of the leakage of gastrointestinal contents, with mediastinitis, septic shock, acute respiratory distress syndrome and death.

Similar results have been shown for colorectal anastomoses. So, a good microcirculatory blood flow around the anastomosis could indicate an optimal condition for anastomotic healing. Or the other way around, a bad microcirculatory blood flow could lead the surgeon to rethink the planned anastomosis.

Objectives: To assess the association of intraoperative flux measurement with postoperative outcome of patients undergoing major abdominal surgery.

Trial design: Prospective observational study. Flux measurement will be carried out using the moorVMS-LDF DUAL CHANNEL Laser Doppler Blood Flow system. The flux probe will be applied on the respective organs (i.e. esophagus, stomach, liver, pancreas, colon, rectum) and measurements will be documented after a stable signal has been obtained.

Laser Doppler measurement allows realtime and continuous monitoring suitable for the investigation of the gastrointestinal microcirculation. Light generated by a laser diode penetrates the tissue, where it is reflected by circulating blood cells. This reflected light is returned via an optical fibre to a photodetector and transformed into an electrical signal, which is proportional to the number of blood cells moving in the measured volume multiplied by the mean velocity of the cells, and is referred to as the blood flux expressed as perfusion units (PU).

Each measurement represents the mean value (PU) of a stable perfusion over a 1-min period without motion artefacts.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective major abdominal surgery including

  * Liver resection
  * Esophageal resection
  * Gastric resection
  * Colon/rectal resection
  * Pancreatic resection

Exclusion Criteria:

* Expected lack of compliance
* Impaired mental state or language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery of liver, stomach, colon/rectum, esophagus, pancreas
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2015-11-18 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-02 (Actual)

PRIMARY OUTCOMES:
Perioperative morbidity | 90 days after resection

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Reißfelder, MD, Principal Investigator — Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany
Locations (1):
- Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, TU Dresden, Germany, Dresden, Saxony, Germany